CLINICAL TRIAL: NCT03357094
Title: Pulmonary Ventilation/Perfusion Imaging With SPECT/CT for the Prediction of Postoperative Residual Pulmonary Function in Patients With Primary Lung Cancer: A Multi-center Clinical Study
Brief Title: Pulmonary Ventilation/Perfusion Imaging for the Prediction of Postoperative Residual Pulmonary Function
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Tongren Hospital (Other)
Collaborators: The First Affiliated Hospital of Zhengzhou University (Other); West China Hospital (Other); Hebei Medical University Fourth Hospital (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); Henan Cancer Hospital (Other Government); Zhejiang Tumor Hospital (Other); RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: tr12345
Record Dates: First submitted 2017-11-23; First posted 2017-11-29 (Actual); Last update posted 2017-11-29 (Actual); Status verified 2017-10

CONDITIONS: Lung Neoplasms
Keywords: Pulmonary ventilation; Pulmonary perfusion; Single Photon Emission Computed Tomography
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Lung cancer is one of the most common malignant tumors in the world and with the highest incidence in China. Surgery is the most effective therapeutic method for primary lung cancer. Accurate prediction of residual postoperative pulmonary function in patients, especially those with borderline pulmonary function, is crucial for proper qualification for surgery. According to the 3rd American College of Chest Physicians(ACCP) evidence-based clinical practice guideline (2013), both predictive postoperative (ppo) FEV1.0% and ppoDLCO% are greater than 60% predicted are required as a first standard of lobectomy for patients with primary lung cancer. And, according to the British Thoracic Society (BTS) guideline, patients with ppoFEV1.0% and ppoDLco% less than 40% have high a risk for surgery. Pulmonary ventilation / perfusion SPECT/CT has recently become available for prediction of lung function, and it can be used to forecast pulmonary function in consideration of the pulmonary circulation as well as effective residual lung function. Traditionally, prediction of postoperative lung function was based on planar method in anterior and posterior projections of lung scintigraphy. However, SPECT/CT enables measurement of ventilation / perfusion uptake in each lobe of the lungs in a three dimensional way, which may avoid underestimating ppoFEV1.0% and provide confidence in suggesting lobectomy or pneumonectomy.

This experiment is intended to explore the use of Q.lung, a volume-based software to semi-quantitatively calculate pulmonary ventilation/perfusion functional uptake and volume by SPECT/CT. We hope it can get a more accurate prediction of postoperative residual pulmonary function to provide better management for clinical surgery.

DETAILED DESCRIPTION:
1. Newly diagnosed and pre-therapeutic patients with primary lung cancer
2. Study sample: the optimal study sample is expected to be >50 cases
3. Inclusion criteria: age 30-80 years old; newly diagnosis of primary lung cancer with radiological or pathological evidence; SPECT/CT scan was performed before surgery; written and informed consent with signature before the study
4. Exclusion criteria: with other tumor in addition to primary lung caner; receive surgery prior to SPECT/CT scan; failed to complete preoperative and postoperative pulmonary function tests; failed to perform scans; pregnancy, lactation, and impaired renal or liver function; poorly controlled diabetes; poor compliance; contrary to the standard operating procedures; not suitable for clinical trials (for example with mental illness);

Study protocol:

1. Examination time

1. Preoperative lung function test was performed within a month prior to surgery
2. Preoperative pulmonary ventilation/perfusion SPECT/CT were performed within a month prior to surgery
3. Postoperative pulmonary function test as well as follow-up were performed within three months after surgery 2. Pulmonary function test including but not limited to: forced expiratory volume in 1s(FEV1), diffusing capacity carbon monoxide(DLCO), forced vital capacity(FVC), maximal voluntary ventilation (MVV), peak expiratory flow(PEFR), vital capacity(VC), total lung capacity(TLC) 3. Pulmonary ventilation/perfusion SPECT/CT imaging: acquisition protocol according to EANM guidelines for ventilation/perfusion scintigraphy. Part 1. Using Technegas for ventilation imaging and 99mTc-MAA for perfusion imaging.

4. Image analysis：

1. Ventilation / perfusion SPECT/CT data were registered, processed and reconstructed in GE Xeleris Workstation, quantitative measurements were using Q.lung software.
2. Results including ventilation / perfusion uptake and volume (in counts and mL and respective percentage) of each pulmonary lobar.

5. Data analysis:

1. Predicted postoperative FEV1 (as well as other pulmonary function values) were calculated according to the following formula:

   FEV1 fore-v = FEV1 pre × (1- Volume%); FEV1 fore-cv = FEV1 pre × (1- Counts%v); FEV1 fore-cp = FEV1 pre × (1- Counts%p).

   *fore-v represents predicted postoperative value using volume; fore-cv represents predicted postoperative value using ventilation uptake; fore-cp represents predicted postoperative value using perfusion uptake; pre represents preoperative pulmonary test value.
2. A graphical method of the Bland-Altman plot was used to compare FEV1 (as well as other pulmonary function values) obtained from predictions and post-operative measurements (with certain systematic and random errors). Intervals of agreement were drawn as the mean difference between predicted and measured values plus and minus 1.96 times the standard deviation of the differences. Strength of linear relationship between predicted and measured FEV1 values was quantified by the Pearson correlation coefficients with significance based on t-statistics. P < 0.05 is statistically significant.

ELIGIBILITY:
Inclusion criteria: age 30-80 years old; newly diagnosis of primary lung cancer with radiological or pathological evidence; SPECT/CT scan was performed before surgery; written and informed consent with signature before the study.

Exclusion criteria: with other tumor in addition to primary lung caner; receive surgery prior to SPECT/CT scan; failed to complete preoperative and postoperative pulmonary function tests; failed to perform scans; pregnancy, lactation, and impaired renal or liver function; poorly controlled diabetes; poor compliance; contrary to the standard operating procedures; not suitable for clinical trials (for example with mental illness);

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed and pre-therapeutic patients with primary lung cancer.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-09-30 (Actual); Primary Completion 2018-11-01 (Estimated); Study Completion 2019-11-01 (Estimated)

PRIMARY OUTCOMES:
compare actual postoperative lung function values to predicted values using residual pulmonary lobar volume by SPECT/CT | 1 month
  using pulmonary lobar volume to calculate predicted postoperative pulmonary test values and compare them with actual postoperative values.
compare actual postoperative lung function values to predicted values using residual ventilation uptake by SPECT/CT | 1 month
  using ventilation uptake (in counts) to calculate predicted postoperative pulmonary test values and compare them with actual postoperative values.
compare actual postoperative lung function values to predicted values using residual perfusion uptake by SPECT/CT | 1 month
  using perfusion uptake (in counts) to calculate predicted postoperative pulmonary test values and compare them with actual postoperative values.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongren Hospital, Beijing, Beijing Municipality, China